CLINICAL TRIAL: NCT06792045
Title: Tongue Motor Functions Assessment As a Screening Tool for Obstructive Sleep Disordered Breathing in Children
Brief Title: Prediction of Tongue Base Obstruction During Sleep
Acronym: PTOS
Status: Not yet recruiting | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, William Poncin, Principal Investigator, Professor, Université Catholique de Louvain
Other Study IDs: PTOS
Record Dates: First submitted 2024-12-22; First posted 2025-01-24 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Obstructive Sleep Disordered Breathing
Keywords: obstructive sleep disordered breathing; pediatrics; sleep; obstructive sleep apnea; snoring; tongue
MeSH Terms: conditions — Sleep Apnea, Obstructive; Snoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children with obstructive sleep disordered breathing
  Interventions: Other: Physiotherapist assessment; Other: ENT assessment; Diagnostic Test: Drug-Induced Sleep Endoscopy

INTERVENTIONS:
Other: Physiotherapist assessment — * Tongue motor skills (Tongue pressures and tongue mobility, assessed through the Iowa Oral Performance Instrument and the Motricité Bucco-Linguo-Faciale tongue subscore, respectively)
  * Tongue restriction of mobility due to its frenulum (assessed through the Quick Tongue-Tie assessment tool)
  * Breathing Pattern (questionnaire from Abreu RR, Rocha RL, Lamounier JA, Guerra AF. Etiology, clinical manifestations and concurrent findings in mouth-breathing children. J Pediatr (Rio J). 2008;84(6):529-535.).
Other: ENT assessment — Data from the ENT appointment will be collected (e.g., sex, height, weight)
Diagnostic Test: Drug-Induced Sleep Endoscopy — A Drug-Induced Sleep Endoscopy will be performed, recorded, and evaluated by two blinded raters using the IPSES scale.

SUMMARY:
This study investigates the hypothesis that, in children, tongue motor functions can predict both the anatomical site and the degree of upper airway obstruction contributing to obstructive sleep-disordered breathing.

DETAILED DESCRIPTION:
Patients will be enrolled during their visit to the ENT physician. Subsequently, their tongue motor functions will be assessed during their pre-surgical appointment. Finally, they will undergo a drug-induced sleep endoscopy prior to their surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 and 17 years old
* Medical diagnosis of obstructive sleep-disordered breathing requiring surgical removal of tonsils (partial or total) and/or adenoids
* Positive Pediatric Sleep Questionnaire (8 or more positive responses)
* Eligibility for surgical intervention

Exclusion Criteria:

* Neurological, cardiac, or respiratory comorbidity other than obstructive sleep-disordered breathing
* Previous surgery of the upper airway or oral cavity
* History of or current head or neck cancer
* Cranial, upper airway, or oral cavity malformation
* Contraindication to performing endoscopy

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will be recruited during ENT consultations.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Extent of tongue base obstruction | During the planned surgery
  Evaluated through the IPSES scoring during a Drug Induced Sleep Endoscopy (DISE)

SECONDARY OUTCOMES:
Breathing pattern | During the pre-surgical appointment
  Presence or absence of mouth breathing will be assessed with the mouth breathing questionnaire from Abreu et al. (2018).
Tongue mobility (MBLF score) | During the pre-surgical appointment
  Assessed through the Motricité Bucco-Linguo-Faciale (MBLF) tongue test score
Tongue pressures (kPa) | During the pre-surgical appointment
  Tongue pressures will be measured with the Iowa Oral Performance Instrument (IOPI), in kPa, during a protrusion, an elevation, and a swallowing task.
Tongue mobility restriction due to its frenulum ratio (%) | During the pre-surgical appointment
  The ratio between the maximal comfortable mouth opening, with the tongue tip to the incisive papilla, and the maximal comfortable mouth opening, will be computed.

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No